CLINICAL TRIAL: NCT02081339
Title: Cohort Study of the Clinical Course of Macular Diseases in Japanese Patients
Brief Title: Cohort Study of the Clinical Course of Macular Diseases in Japanese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Nagahisa Yoshimura, Professor, Kyoto University, Graduate School of Medicine
Other Study IDs: E2038
Record Dates: First submitted 2014-01-22; First posted 2014-03-07 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Macular Disease
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; aflibercept; pegaptanib; Verteporfin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Macular diseases: ranibizumab, intravitreal injections, 0.5mg, monthly or less aflibercept,intravitreal injections, 2.0mg, monthly or less pegaptanib, intravitreal injections, 0.3mg, every 6-week pars plana vitrectomy, once verteporphin, iv, 6mg/㎡
  Interventions: Drug: ranibizumab, aflibercept, pegaptanib, verteporphin

INTERVENTIONS:
Drug: ranibizumab, aflibercept, pegaptanib, verteporphin

SUMMARY:
Recent clinical introduction of anti-vascular endothelial growth factor agents may change the clinical course of macular diseases, including age-related macular degeneration (AMD), polypoidal choroidal vasculopathy (PCV), retinal angiomatous proliferation (RAP), central serous chorioretinopathy (CSC), myopic choroidal neovascularization (CNV), retinal vein occlusion (RVO), diabetic macular edema (DME), and so forth.

Patients with such macular diseases are registered and and are followed up for 5 years with appropriate treatment for each patient. By the analysis of the correlation between initial examinations and final visual acuity, factors associated with good visual prognosis will be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visit Department of Ophthalmology Kyoto University Hospital with macular diseases.
* Patients who are agreed with the participation of this study.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who visit Department of Ophthalmology Kyoto University Hospital with macular diseases.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-03; Primary Completion 2022-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Initial factors associated with visual prognosis in each macular disease | Five years after the registration

SECONDARY OUTCOMES:
The difference in the visual prognosis depending on the treatments in each macular diseases | Five years after the registration

OTHER OUTCOMES:
The change in visual acuity in each macular diseases. | Five years after the registration.

CONTACTS AND LOCATIONS:
Overall Officials: Nagahisa Yoshimura, MD, Study Chair — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University Graduate School of Medicine, Kyoto, Kyoto, Japan